CLINICAL TRIAL: NCT05356364
Title: Improving Negative Stressful Perseverations in Insomnia to Revitalize Expecting Moms (INSPIRE)
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David Kalmbach, Assistant Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34MH130562 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-05-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-05

CONDITIONS: Insomnia; Depression
Keywords: Pregnancy; Postpartum; Telemedicine; Cognitive arousal; Insomnia; Depression; Mindfulness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Cognitive Behavioral Therapy; Sleep

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perinatal Understanding of Mindful Awareness for Sleep (PUMAS) (Active Comparator): PUMAS combines behavioral sleep strategies with elements from mindfulness-based interventions, and is tailored specifically to meet the unique needs of pregnant women. Behavioral sleep strategies include sleep restriction and stimulus control. Mindfulness elements include guided meditations and engaging in mindful activities. PUMAS consists of 6 60-minute sessions with a therapist along with self-monitoring with sleep diaries. All sessions are delivered via telemedicine during pregnancy.
  Interventions: Behavioral: Perinatal Understanding of Mindful Awareness for Sleep (PUMAS)
- Cognitive Behavioral Therapy for Insomnia (CBTI) (Active Comparator): CBTI combines behavioral sleep strategies with cognitive therapy. It is the first-line treatment for insomnia as recommended by the American College of Physicians and the American Academy of Sleep Medicine. Behavioral sleep strategies include sleep restriction and stimulus control. Cognitive therapy includes scheduled worry time and challenging dysfunctional beliefs about sleep. CBTI consists of 6 60-minute sessions with a therapist along with self-monitoring with sleep diaries. All sessions are delivered via telemedicine during pregnancy.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTI)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBTI) — cognitive and behavioral treatment for perinatal insomnia.
  Arms: Cognitive Behavioral Therapy for Insomnia (CBTI)
Behavioral: Perinatal Understanding of Mindful Awareness for Sleep (PUMAS) — Mindfulness and behavioral based therapy for perinatal insomnia.
  Arms: Perinatal Understanding of Mindful Awareness for Sleep (PUMAS)

SUMMARY:
Nearly half of women develop insomnia during pregnancy, which is associated with increased risk for developing perinatal depression. The purpose of this research is to evaluate the implementability and effectiveness of a mindfulness-based therapy for insomnia relative to cognitive-behavioral therapy for insomnia in pregnant women with insomnia and comorbid depression. The investigators aim to examine whether a mindfulness-based intervention effectiveness reduces symptoms of insomnia and comorbid depression.

DETAILED DESCRIPTION:
The investigators will conduct a pilot hybrid type 1 effectiveness-implementation randomized controlled trial (RCT) wherein 100 pregnant women with DSM-5 insomnia disorder and comorbid depression (Edinburgh Postnatal Depression Scale ≥ 10) are randomized to a mindfulness-based intervention--Perinatal Understanding of Mindful Awareness for Sleep (PUMAS)--or Cognitive Behavioral Therapy for Insomnia (CBTI). Patients will be recruited from women's health clinics across Henry Ford Health in Metro Detroit including underserved women, serving as real-world implementation. Per clinic operations since the pandemic, therapies will be via telemedicine to meet patient expectations. Study outcomes will be assessed before and after treatment, then across the first postpartum year.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy, gestational week 14-31.
2. DSM-5 Insomnia Disorder (acute or chronic).
3. Insomnia Severity Index (ISI) score ≥ 11.
4. Edinburgh Postnatal Depression Scale (EPDS) score ≥ 10.
5. Ensure adequate sleep opportunity.
6. Age ≥ 18, English-speaking.
7. Reliable internet access (treatment, assessments)

Exclusion Criteria:

1. High risk pregnancy (age >40y, pre-eclampsia, any condition deemed serious risk to mother/fetus; hypertension and diabetes allowed).
2. Active suicidal intent (ideation is allowed).
3. Night or rotating shift work.
4. Epworth Sleepiness Scale>15 (Excessive sleepiness)
5. Health condition unsafe for sleep restriction (bipolar, epilepsy, etc.).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant women are eligible to participate in this trial.
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Comparative effectiveness between PUMAS and CBTI on acute insomnia effects. | The investigators will examine change in ISI scores from Pretreatment Baseline to Posttreatment, the latter will occur 6-9 weeks after Baseline.
  The Insomnia Severity Index (ISI) is a commonly used self-report measure of insomnia symptoms that has been validated in a perinatal sample. The ISI scores range from 0-28 with higher scores indicating greater insomnia severity.
Comparative effectiveness between PUMAS and CBTI on postpartum insomnia effects. | The investigators will examine changes in ISI scores across the first postnatal year, which will be assessed at 3, 6, 9, and 12 months postpartum..
  The Insomnia Severity Index (ISI) is a commonly used self-report measure of insomnia symptoms that has been validated in a perinatal sample. The ISI scores range from 0-28 with higher scores indicating greater insomnia severity.

SECONDARY OUTCOMES:
Comparative effectiveness between PUMAS and CBTI on acute depression effects. | The investigators will examine change in EPDS scores from Pretreatment Baseline to Posttreatment, the latter will occur 6-9 weeks after Baseline.
  The Edinburgh Postnatal Depression Scale (EPDS) is the most widely used depression measure in both pregnant and postnatal women. It is validated for use in clinical trials. The EPDS scores range from 0-30 with higher scores indicating greater depression severity.
Comparative effectiveness between PUMAS and CBTI on postpartum depression effects. | The investigators will examine changes in EPDS scores across the first postnatal year, which will be assessed at 3, 6, 9, and 12 months postpartum.
  The Edinburgh Postnatal Depression Scale (EPDS) is the most widely used depression measure in both pregnant and postnatal women. It is validated for use in clinical trials. The EPDS scores range from 0-30 with higher scores indicating greater depression severity.
Comparative effectiveness between PUMAS and CBTI on acute cognitive arousal effects. | The investigators will examine change in PSASC scores from Pretreatment Baseline to Posttreatment, the latter will occur 6-9 weeks after Baseline.
  The Pre-Sleep Arousal Scale's Cognitive factor (PSASC) is a self-report measure of nocturnal cognitive arousal that has been validated in the perinatal population. Scores range form 8-40 with higher scores indicating greater nighttime cognitive arousal.
Comparative effectiveness between PUMAS and CBTI on postpartum cognitive arousal effects. | The investigators will examine changes in PSASC scores across the first postnatal year, which will be assessed at 3, 6, 9, and 12 months postpartum.
  The Pre-Sleep Arousal Scale's Cognitive factor (PSASC) is a self-report measure of nocturnal cognitive arousal that has been validated in the perinatal population. Scores range form 8-40 with higher scores indicating greater nighttime cognitive arousal.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No